CLINICAL TRIAL: NCT06505837
Title: Open-Label, Randomized, Phase III Clinical Study Comparing the Pharmacokinetic Profile, Efficacy, and Safety of JS001sc and JS001 in Combination With Standard Chemotherapy as First-Line Treatment for Recurrent Metastatic Non-Squamous Non Small Cell Lung Cancer
Brief Title: JS001sc or JS001 Plus Chemotherapy is Indicated for Relapsed or Metastatic First-Line Non-Squamous Non Small Cell Lung Cancer（NSCLC）
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS001sc-002-III-NSCLC
Record Dates: First submitted 2024-05-19; First posted 2024-07-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Metastatic Non-Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — Injections, Subcutaneous; Pemetrexed; Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Parallel
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1:JS001sc (360mg Subcutaneous injection) and pemetrexed/platinum-containing chemotherapy (Experimental)
  Interventions: Drug: JS001sc (360mg Subcutaneous injection) and pemetrexed/platinum-containing chemotherapy
- Arm 2:JS001 (240mg intravenous infusion) and pemetrexed/platinum-containing chemotherapy (Active Comparator)
  Interventions: Drug: JS001 (240mg intravenous infusion) and pemetrexed/platinum-containing chemotherapy

INTERVENTIONS:
Drug: JS001sc (360mg Subcutaneous injection) and pemetrexed/platinum-containing chemotherapy — The combination therapy of JS001sc and pemetrexed/platinum lasted for 4 cycles, after which subjects who did not progress continued to receive JS001sc and pemetrexed maintenance therapy, and the cumulative treatment of JS001sc did not exceed 35 cycles (Each cycle is 21 days).
  Arms: Arm1:JS001sc (360mg Subcutaneous injection) and pemetrexed/platinum-containing chemotherapy
Drug: JS001 (240mg intravenous infusion) and pemetrexed/platinum-containing chemotherapy — The combination therapy of JS001 and pemetrexed/platinum lasted for 4 cycles, after which subjects who did not progress continued to receive JS001 and pemetrexed maintenance therapy, and the cumulative treatment of JS001 did not exceed 35 cycles (Each cycle is 21 days).
  Arms: Arm 2:JS001 (240mg intravenous infusion) and pemetrexed/platinum-containing chemotherapy

SUMMARY:
This is a multicenter, open-Lable, randomized, phase III clinical study to compare the pharmacokinetic profile, efficacy, and safety of Toripalimab injection (subcutaneous) (JS001sc) and Toripalimab injection (JS001) in combination with standard chemotherapy as first-line treatment for recurrent or metastatic Non-Squamous Non small cell lung cancer

DETAILED DESCRIPTION:
This study adopted a randomized, open-label, positive control, multicenter, phase III clinical research design. It selected patients with recurrent or metastatic non-squamous NSCLC who did not have sensitive EGFR mutations or ALK fusions. A total of 356 patients (increased to 395 according to the recommendation of the Data Monitoring Committee) were planned to be enrolled. They would be randomly assigned to one of the following two treatment groups at a ratio of 1:1:

Group A: JS001sc+ platinum-based chemotherapy

JS001sc, 360 mg, was administered subcutaneously (SC) once every 3 weeks (Q3W).

Chemotherapy: pemetrexed + carboplatin/cisplatin, Q3W, up to 4 cycles, non-progressive subjects pemetrexed monotherapy maintenance therapy.

Group B: JS001+ platinum-based chemotherapy

JS001, 240 mg, IV, Q3W.

Chemotherapy: pemetrexed + carboplatin/cisplatin, Q3W, up to 4 cycles, non-progressive subjects pemetrexed monotherapy maintenance therapy.

Both groups were treated until treatment termination criteria were met.

This study was divided into screening, treatment and follow-up periods.

Screening period

After signing the Informed consent form (ICF), the subjects entered the study screening period. The screening period was up to 28 days, and subjects who met all inclusion criteria and did not meet any exclusion criteria entered the study treatment period.

Period of treatment

Tests and evaluations should be completed before each dose. Subjects were assigned to receive JS001sc or JS001 combined with pemetrexed plus carboplatin/cisplatin chemotherapy until the criteria for treatment discontinuation were met. Patients with progressive disease (PD) according to RECIST v1.1 criteria at the first evaluation were allowed to continue treatment until the criteria for discontinuation of treatment were met after discussion with the sponsor and with the investigator's judgment that the patient was clinically stable and could potentially continue to benefit.

During the study, the efficacy will be evaluated per RECIST v1.1 criteria.

Protocol efficacy and safety assessments should be completed according to the Evaluation Schedule (SoA).

Follow-up period

The safety follow-ups were 30 days (±7 days) and 90 days (±7 days) after the last study dose or before starting a new antitumor therapy, whichever occurred first.

Survival follow-up was performed every 30 days (±7 days) from the last dose of medication until death, loss to follow-up, withdrawal of consent, or termination of the study by the sponsor.

ELIGIBILITY:
Inclusion criteria：

1. Age ≥18 years at the time of signing informed consent, both male and female.
2. Histologically or cytologically confirmed relapsed or metastatic non-squamous NSCLC.
3. A test report confirming the absence of EGFR sensitive mutations and ALK fusions (local laboratory reports are acceptable, but the tests must be well-validated and either pass external quality assessment or be qualified for molecular pathology diagnosis/gene testing or approved by NMPA).
4. No prior systemic anti-tumor therapy for advanced or metastatic non-squamous NSCLC. Subjects who have received adjuvant therapy or neoadjuvant therapy (chemotherapy, radiotherapy, or other treatments) for recurrent non-squamous NSCLC can be enrolled if the interval between the last treatment and recurrence is more than 6 months.
5. Subject has at least 1 measurable lesion according to RECIST v1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
7. Expected survival ≥ 12 weeks.
8. The function of vital organs meets the following requirements (Note: no blood components and hematopoietic growth factors are allowed to be used within 14 days before screening);

   1. Absolute neutrophil count (ANC) ≥1.5×109/L；
   2. Platelet ≥ 100×109/L;
   3. Hemoglobin ≥9 g/dL;
   4. Bilirubin ≤1.5× upper limit of normal (ULN);
   5. Alanine aminotransferase (ALT) ≤ 2.5× ULN, aspartate aminotransferase (AST) ≤ 2.5× ULN;
   6. Creatinine clearance (CrCL) ≥ 60 mL/min (cisplatin) or CrCL ≥50 mL/min (carboplatin) (Cockcroft-Gault formula);
   7. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, International normalized ratio (INR) ≤ 1.5 (for prophylactic anticoagulation at stable doses, drug-specific monitoring requirements are acceptable beyond this range)；
9. Female subjects who are capable of reproduction, as well as male subjects whose partners are of childbearing age (as listed in Appendix 5), are required to use an effective form of contraception during the study treatment period and for at least 6 months after the last treatment (as stated in Appendix 7)；
10. Voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up plan；

Exclusion criteria：

1. Concomitant study disease states of：

   1. Histological or cytological pathology of the tumor confirmed with small cell lung cancer component or sarcomatoid lesion, or squamous cell carcinoma component >10%;
   2. Patients with known meningeal metastasis; patients with symptomatic brain metastases; patients with asymptomatic brain metastases, who have been evaluated by the investigators as stable can be enrolled, including: 1) Those who have maintained stability after receiving radiotherapy for brain metastases, and the stability criteria need to meet all of the following conditions: no symptoms related to brain metastases, at least 7 days before the administration of the study drug, no disease progression was found in the imaging examination after the brain metastasis treatment compared to the imaging examination before the treatment (at least a 4-week interval); 2) Those without local treatment for asymptomatic brain metastases, and need to meet all of the following conditions: no use of corticosteroids or other drugs to control symptoms related to brain metastases, no long diameter of any brain metastasis lesion ≥ 1 cm, no metastasis in the midbrain, pons, medulla oblongata, cerebellum or spinal cord, and no history of intracranial hemorrhage in the past;
   3. Uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage (once a month or more frequently); subjects with stable symptoms after drainage for at least two weeks can be enrolled;
   4. Spinal cord compression that has not been treated surgically and/or radiotherapeutically, or those diagnosed with spinal cord compression in the past who have no clinical evidence showing disease stability ≥ 4 weeks before enrollment;
   5. Known to have other existing standard first-line treatment-driven gene mutations, including but not limited to: ROS1 fusion, BRAF V600 mutation, MET14 exon skipping mutation, RET fusion;2. Have received any of the following treatments；
2. Have received any of the following treatments:

   1. Received local small-area radiotherapy (such as palliative radiotherapy for bone metastases) within 14 days prior to the first study drug administration;
   2. Prior immune-mediated therapy, including but not limited to anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy (or any other antibodies acting on T cell synergistic stimulation or checkpoint pathways such as IDO, IL-2R, GITR);
   3. Receipt of any investigational drug within 4 weeks or 5 half-lives prior to the first dose of study drug, whichever is shorter;
   4. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study, or the subject is in the follow-up period of the interventional clinical study;
   5. Systemic therapy with corticosteroids (> 10 mg prednisone equivalent dose per day) or other immunosuppressants within 2 weeks prior to the first dose of study drug. Inhaled or topical corticosteroids are permitted. Receipt of short-term corticosteroids (such as pre-intravenous contrast) within 2 weeks prior to the first dose of study drug is permitted;
   6. Subjects who have received proprietary Chinese medicines or immunomodulatory drugs with anti-tumor indications (thymus peptide, interferon, interleukin, etc.) within 2 weeks before the first dose of study drug, or who need to continue to receive these drugs during the study;
   7. Those who have been vaccinated with anti-tumor vaccines or have received live vaccines within 4 weeks before the first dose of study drug;
   8. Major surgery or severe trauma within 4 weeks prior to the first use of study drug；
3. Toxicity from previous anti-tumor therapy has not recovered to ≤ CTCAE grade 1 (except for toxicity judged by the investigator to have no safety risk);
4. Known hypersensitivity to any of the study treatments and their excipients;
5. Unable or unwilling to use folic acid or vitamin B12 injection;
6. Active autoimmune disease, history of autoimmune disease (including but not limited to interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism); except for:

   1. Subjects with vitiligo or cured childhood asthma/allergies that do not require any intervention after adulthood;
   2. Subjects with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone;
   3. Subjects on stable doses of insulin for the treatment of type I diabetes mellitus;
   4. Subjects with well-controlled hyperthyroidism after adequate treatment；
7. Have a history of immunodeficiency, including a positive HIV test, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
8. Severe infection (CTCAE> grade 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, infection comorbidities, etc., active lung inflammation on baseline chest imaging, symptoms and signs of infection within 2 weeks prior to the first dose of the study drug requiring oral or intravenous antibiotic treatment (except for prophylactic antibiotic use);
9. Confirmed or suspected history of interstitial lung disease or idiopathic pulmonary fibrosis, drug-induced pneumonitis, idiopathic pneumonitis, or other moderate to severe pulmonary diseases that seriously affect lung function (except for ≤ grade 1 radiation pneumonitis);
10. Subjects with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or subjects with a history of active pulmonary tuberculosis infection more than 1 year ago but without formal treatment;
11. Presence of active hepatitis B (hepatitis B virus surface antigen (HBsAg) positive with HBV DNA ≥500 IU/mL), hepatitis C (hepatitis C antibody positive, and HCV-RNA above the lower limit of detection of the analytical method);
12. Diagnosis of any other malignancy prior to the first dose of study drug within 5 years, with the exception of malignancies with low risk of metastasis (5-year survival rate >90%), such as adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or adequately treated localized prostate cancer;
13. Pregnant or lactating women;
14. Uncontrolled concurrent diseases, including but not limited to: symptomatic congestive heart failure, left ventricular ejection fraction (LVEF) < 50%, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, major epileptic seizures, superior vena cava syndrome, or other conditions that may affect study compliance, significantly increase the risk of adverse events, or impair the ability of subjects to provide written informed consent; such as mental disorders/societal conditions；
15. As judged by the investigator, the subject has other factors that may lead to the forced termination of the study, such as other serious diseases (including mental illnesses) requiring concomitant treatment, serious abnormalities in laboratory test values, and/or family or social factors that may affect the safety of the subject or the collection of experimental data；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Observed serum Ctrough at Cycle 1 | the end of Cycle 1 (Each cycle is 21 days)
  Measured valley concentration at the end of cycle 1 (Ctrough)
Model-predicted area under the concentration-time curve(AUC) from 0 to 21 days at Cycle 1 | the end of Cycle 1 (Each cycle is 21 days)
  The area under the drug time curve of cycle 1 simulated by a population pharmacokinetic model

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 2years
  Comparison of Objective response rate (ORR) between JS001sc and JS001 in first-line patients with relapsed or metastatic non-squamous NSCLC
Progression-free survival (PFS) | up to 2years
  Comparison of first-line Progression-free survival (PFS) between JS001sc and JS001 in patients treated with relapsed or metastatic non-squamous NSCLC
6-month progression-free survival(PFS) rate | up to 6-month
  The 6-month progression-free survival(PFS) rate in first-line patients treated with relapsed or metastatic non-squamous NSCLC was compared between JS001sc and JS001
Disease control rate (DCR) | up to 2years
  Comparison of first-line Disease control rate (DCR) between JS001sc and JS001 in patients with relapsed or metastatic non-squamous NSCLC
Duration of response (DoR) | up to 2years
  Comparison of first-line Duration of response (DoR) between JS001sc and JS001 in patients treated with relapsed or metastatic non-squamous NSCLC
Safety: adverse events (AEs) | up to 2years
  The safety of JS001sc and JS001 as first-line treatment in subjects with relapsed or metastatic non-squamous-scale NSCLC was compared by adverse event rate (percentage of participants with treaty-related adverse events assessed by CTCAEv5.0) and abnormal laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Wang, doctorate, Study Director — Medical director
Locations (1):
- Hunan Cancer Hospital, Changshang, Hunan, China

IPD SHARING:
Plan to Share IPD: No